CLINICAL TRIAL: NCT03077867
Title: Comparison of Histological and Radiographic Evidence After Sinus Lift With Synthetic Nano-hydroxyapatite and Inorganic Bovine Bone.
Brief Title: Comparison Synthetic Hydroxyapatite and Inorganic Bovine Bone in Sinus Floor Elevation
Acronym: SYNBIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Piezosurgery Academy (Other)
Collaborators: University of Trieste (Other)
Responsible Party: Principal Investigator, Mr. Claudio Stacchi, DDS, MSc, President of the International Piezosurgery Academy, International Piezosurgery Academy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SINBYO
Record Dates: First submitted 2017-01-25; First posted 2017-03-13 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Alveolar Bone Loss
Keywords: sinus lift; synthetic hydroxyapatite; bone graft
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Sinus Floor Augmentation; Bone Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- test HA (Experimental): synthetic hydroxyapatite alone sinus floor augmentation with bone graft
  Interventions: Procedure: sinus floor augmentation with bone graft
- test HA vicryl (Experimental): synthetic hydroxyapatite mixed with polylactic-polyglycolic acid sinus floor augmentation with bone graft
  Interventions: Procedure: sinus floor augmentation with bone graft
- test HA-PRF (Experimental): synthetic hydroxyapatite mixed with i-PRF sinus floor augmentation with bone graft
  Interventions: Procedure: sinus floor augmentation with bone graft
- control (Active Comparator): anorganic bovine bone sinus floor augmentation with bone graft
  Interventions: Procedure: sinus floor augmentation with bone graft

INTERVENTIONS:
Procedure: sinus floor augmentation with bone graft — sinus floor augmentation with lateral approach with bone graft
  Other Names: LASFE

SUMMARY:
This is set as prospective clinical trial to correlate histologically and radiologically the performance of four different bone grafts (synthetic hydroxyapatite alone, synthetic hydroxyapatite mixed with polylactic-polyglycolic acid, synthetic hydroxyapatite with i-PRF and inorganic bone graft) in the sinus floor elevation technique with lateral approach for the treatment of atrophic crests.

DETAILED DESCRIPTION:
SURGICAL PROCEDURE:

After local anesthesia and a large full-thickness mucoperiosteal flap in the area of interest, an osteotomy window on the side wall of the maxillary sinus will be opened using bone scrapers and / or ultrasonic instruments. Will be recorded the time needed for the opening dell'antrostomy and any perforations of the membrane at this stage. The Schneider membrane is then gently elevated with ultrasonic instrumentation and curettes manuals: after testing the integrity of the membrane by means of visual inspection and the Valsalva maneuver, the sealed envelope in which will be indicated to the surgeon the material to be used as a graft will be opened. The biomaterials selected for this study are a synthetic nano-hydroxyapatite (SNHA) (FISIOGRAFT Bone, Italy), to be used either alone, or mixed with a polylactic- polyglycolic copolymer (PLGA) (FISIOGRAFT, Italy), or mixed with autologous platelet derived (i-PRF) and inorganic bovine bone (ABB) (Bio-Oss, Geistlich, Switzerland). After completing the insertion of the biomaterial, the antrostomy will be protected with a resorbable collagen membrane (BioGide, Geistlich, Switzerland) and the flaps will be sutured with a synthetic monofilament.

It will prescribe antibiotics for 6 days (amoxicillin 1 g twice daily or, in allergic patients, clarithromycin 250 mg twice a day) and NSAIDs (ibuprofen 600 mg), as needed. An aerosol treatment with beclomethasone dipropionate and n-acetylcysteine (Fluimucil, Zambon, Italy) will be prescribed at the discretion of the clinician.

POSTOPERATIVE RECALLS:

The sutures will be removed after 10 days and a cone beam computed tomography X-ray will be performed to assess the correct distribution of the graft material and early intercept any accidental leakage of the same in the sinus cavities.

After six months it will proceed to a new radiographic evaluation to assess the resulting regeneration and be able to plan the implant placement.

It will then proceed to the preparation of the sites for the implants using twist-drills. The fixtures are left healed submerged for a period of four months, at the end of which will be connected with the healing screws to start the prosthetic procedures.

After therapy patients will enter a maintenance program with periodic reminders of professional oral hygiene. Patients will be re-evaluated clinically and radiologically after one, three and five years to control the condition of the plants and the stability of the performed regeneration.

ELIGIBILITY:
Inclusion Criteria:

1. indications for intervention of sinus lift with lateral approach to allow the insertion of dental implants, based on careful diagnosis and treatment plan;
2. presence of residual bone crest with a height ≤3 mm on the maxillary sinus, at the level of the implant sites planned;
3. the bone crest must be intact (at least 3 months after the loss / extraction of the element corresponding tooth);

5) patients must be able to examine and understand the study protocol; 6) informed consent.

Exclusion Criteria:

1. acute myocardial infarction within the last six months;
2. uncontrolled bleeding disorders;
3. uncontrolled diabetes (HBA1c> 7.5%);
4. radiation therapy in the district head / neck in the last 24 months;
5. immunocompromised (e.g. HIV infection or chemotherapy in the last three years);
6. current or past treatment with intravenous bisphosphonates;
7. allergy to bovine collagen;
8. psychological or psychiatric diseases;
9. abuse of alcohol or drug use;
10. not controlled periodontal disease;
11. sinus disorders that contraindicate the maxillary sinus lift

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2017-01-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
comparison of histological performance of the bone grafts | 6 months after surgery
  histomorphometric analysis

SECONDARY OUTCOMES:
implant success | 6 months after surgery
  clinical and radiological success of implants inserted in augmented sites
comparison of radiological evidence of the bone grafts | before surgery and 6 months after surgery
  cone beam computed tomography scans of the augmented sinuses

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Stacchi, Dr., Study Director — Piezosurgery Academy
Locations (1):
- Piezosurgery Academy, Parma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farina R, Pramstraller M, Franceschetti G, Pramstraller C, Trombelli L. Alveolar ridge dimensions in maxillary posterior sextants: a retrospective comparative study of dentate and edentulous sites using computerized tomography data. Clin Oral Implants Res. 2011 Oct;22(10):1138-1144. doi: 10.1111/j.1600-0501.2010.02087.x. Epub 2011 Feb 15. PMID 21320169
- [Result] Del Fabbro M, Testori T, Francetti L, Weinstein R. Systematic review of survival rates for implants placed in the grafted maxillary sinus. Int J Periodontics Restorative Dent. 2004 Dec;24(6):565-77. PMID 15626319